CLINICAL TRIAL: NCT02999191
Title: Relative Bioavailability of a BI 1467335 Tablet Compared to a BI 1467335 Oral Solution and the Effect of Food on the Bioavailability of the Tablet Following Oral Administration (a Randomised, Open-label, Single Dose, Three-way Crossover Trial in Healthy Male Subjects)
Brief Title: Relative Bioavailability of BI 1467335 Tablet and Oral Solution, and Food Effect on Tablet in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1386.17; 2016-001534-97 (EudraCT Number)
Record Dates: First submitted 2016-12-19; First posted 2016-12-21 (Estimated); Results first posted 2021-06-07 (Actual); Last update posted 2021-06-07 (Actual); Status verified 2021-05

CONDITIONS: Healthy Volunteers

ARMS (3):
- BI 1467335 (Treatment A) (Experimental): Tablet under fasted conditions
  Interventions: Drug: BI 1467335 (Treatment A)
- BI 1467335 (Treatment B) (Experimental): Oral solution under fasted conditions
  Interventions: Drug: BI 1467335 (Treatment B)
- BI 1467335 (Treatment C) (Experimental): Tablet under fed conditions
  Interventions: Drug: BI 1467335 (Treatment C)

INTERVENTIONS:
Drug: BI 1467335 (Treatment A)
  Arms: BI 1467335 (Treatment A)
Drug: BI 1467335 (Treatment B)
  Arms: BI 1467335 (Treatment B)
Drug: BI 1467335 (Treatment C)
  Arms: BI 1467335 (Treatment C)

SUMMARY:
The primary objective of this trial is to investigate the relative bioavailability of BI 1467335, given as film-coated tablet compared to BI 1467335, given as oral solution. This assessment will be performed under fasted conditions. Furthermore, the effect of food on relative bioavailability of the tablet formulation of BI 1467335 will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects according to the investigators assessment, based on a complete medical history including a physical examination, vital signs (Blood Pressure (BP),Pulse Rate(PR)), 12-lead Electrocardiogram (ECG), and clinical laboratory tests
* Age of 18 to 55 years (incl.)
* Body Mass Index (BMI) of 18.5 to 29.9 kg/m2 (incl.)
* Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice (GCP) and local legislation
* Willingness to comply with contraception requirements. Subjects who are sexually active, must use, with their female partner, adequate contraception throughout the study and until one month after the last administration of trial medication. Adequate methods are:

  * Sexual abstinence or
  * A vasectomy performed at least 1 year prior to screening in combination with a barrier method (condom or diaphragm) or
  * Surgical sterilisation (including bilateral tubal occlusion, hysterectomy or bilateral oophorectomy) of the subjects female partner or
  * The use of condoms, if the female partner uses in addition an adequate contraception method, e.g., intrauterine device (IUD), hormonal contraception (e.g. implants, injectables, combined oral or vaginal contraceptives) that started at least 2 months prior to first drug administration, or barrier method (e.g. diaphragm with spermicide) Unprotected sexual intercourse with a pregnant female partner is not allowed throughout the study and until one month after the last administration of trial medication.

Exclusion Criteria:

* Any finding in the medical examination (including Blood Pressure (BP), Pulse Rate (PR) or Electrocardiogram (ECG) is deviating from normal and judged as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 50 to 90 beats per minute (bpm)
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease judged as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Cholecystectomy and/or surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy and simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* Chronic or relevant acute infections
* History of relevant allergy or hypersensitivity (including allergy to the trial medication or its excipients)
* Use of drugs within 30 days prior to administration of trial medication, if that might reasonably influence the results of the trial (incl. QT/QTc interval prolongation)
* Participation in another trial where an investigational drug has been administered within 60 days prior to planned administration of trial medication or current participation in another trial involving administration of investigational drug
* Smoker (more than 10 cigarettes or 3 cigars or 3 pipes per day)
* Inability to refrain from smoking on specified trial days
* Alcohol abuse (consumption of more than 30 g per day)
* Drug abuse or positive drug screening
* Blood donation of more than 100 mL within 30 days prior to administration of trial medication or intended donation during the trial
* Intention to perform excessive physical activities within 7 days prior to administration of trial medication or during the trial
* Inability to comply with dietary regimen of trial site
* A marked baseline prolongation of QT/QTc interval (such as QTc intervals that are repeatedly greater than 450 ms) or any other relevant ECG finding at screening
* A history of additional risk factors for Torsades de Pointes (such as heart failure, hypokalaemia, or family history of Long QT Syndrome)
* Subject is assessed as unsuitable for inclusion by the investigator, for instance, because considered not able to understand and comply with study requirements, or has a condition that would not allow safe participation in the study

In addition, the following trial-specific exclusion criteria apply:

- Cataract in the medical history

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2017-01-10 (Actual); Primary Completion 2017-03-15 (Actual); Study Completion 2017-04-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- Humanpharmakologisches Zentrum Biberach, Biberach, Germany

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was randomised, open-label, single-dose, three-way crossover trial. 18 subjects entered in the study. 18 subjects were treated in Treatment A: BI 1467335 10 mg tablets, fasted. 18 subjects were treated in Treatment B: BI 1467335 10 mg oral solution, fasted and 17 subjects were treated in Treatment C: BI 1467335 10 mg tablets, fed.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria.
  Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Groups:
- BI 1467335: Tablets, Fasted/Solution, Fasted/Tablets, Fed: The subjects were administered BI 1467335 10 mg [2*5 mg] film-coated tablets orally in the fasted state [Treatment A] in period 1, followed by BI 1467335 10 mg oral solution in the fasted state orally with 240 mL of water after an overnight fast of at least 10 hours [h] [Treatment B] in period 2, then followed by BI 1467335 10 mg [2*5 mg] film-coated tablets orally in the fed state [Treatment C] in period 3. The treatment duration was one day for each treatment [3 single doses], separated by washout phases of at least 21 days.
- BI 1467335: Solution, Fasted/Tablets, Fed/Tablets, Fasted: The subjects were administered BI 1467335 10 mg oral solution in the fasted state orally with 240 mL of water after an overnight fast at least 10h [Treatment B] in period 1, followed by BI 1467335 10 mg [2*5 mg] film-coated tablets orally in the fed state [Treatment C] in period 2, then followed by BI 1467335 10 mg [2*5 mg] film-coated tablets in the fasted state [Treatment A] orally with 240 mL of water after an overnight fast of at least 10h in period 3. The treatment duration was one day for each treatment [3 single doses], separated by washout phases of at least 21 days.
- BI 1467335: Tablets, Fed/Tablets, Fasted/Solution, Fasted: The subjects were administered BI 1467335 10 mg [2*5 mg] film-coated tablets orally in the fed state [Treatment C] in period 1, followed by BI 1467335 10 mg [2*5 mg] film-coated tablets orally in the fasted state [Treatment A] in period 2, then followed by BI 1467335 10 mg oral solution in the fasted state orally with 240 mL of water after an overnight fast of at least 10h [Treatment B] in period 3. The treatment duration was one day for each treatment [3 single doses], separated by washout phases of at least 21 days.
Period: Treatment Period 1 [1 Day]
Arm/Group | BI 1467335: Tablets, Fasted/Solution, Fasted/Tablets, Fed | BI 1467335: Solution, Fasted/Tablets, Fed/Tablets, Fasted | BI 1467335: Tablets, Fed/Tablets, Fasted/Solution, Fasted
Started | 6 | 6 | 6
Completed | 6 | 6 | 6
Not Completed | 0 | 0 | 0
Period: Wash-out Period 1 [21 Days]
Arm/Group | BI 1467335: Tablets, Fasted/Solution, Fasted/Tablets, Fed | BI 1467335: Solution, Fasted/Tablets, Fed/Tablets, Fasted | BI 1467335: Tablets, Fed/Tablets, Fasted/Solution, Fasted
Started | 6 | 6 | 6
Completed | 6 | 5 | 6
Not Completed | 0 | 1 | 0
Not completed — Adverse Event | 0 | 1 | 0
Period: Treatment Period 2 [1 Day]
Arm/Group | BI 1467335: Tablets, Fasted/Solution, Fasted/Tablets, Fed | BI 1467335: Solution, Fasted/Tablets, Fed/Tablets, Fasted | BI 1467335: Tablets, Fed/Tablets, Fasted/Solution, Fasted
Started | 6 | 5 | 6
Completed | 6 | 5 | 6
Not Completed | 0 | 0 | 0
Period: Wash-out Period 2 [21 Days]
Arm/Group | BI 1467335: Tablets, Fasted/Solution, Fasted/Tablets, Fed | BI 1467335: Solution, Fasted/Tablets, Fed/Tablets, Fasted | BI 1467335: Tablets, Fed/Tablets, Fasted/Solution, Fasted
Started | 6 | 5 | 6
Completed | 6 | 5 | 6
Not Completed | 0 | 0 | 0
Period: Treatment Period 3 [1 Day]
Arm/Group | BI 1467335: Tablets, Fasted/Solution, Fasted/Tablets, Fed | BI 1467335: Solution, Fasted/Tablets, Fed/Tablets, Fasted | BI 1467335: Tablets, Fed/Tablets, Fasted/Solution, Fasted
Started | 6 | 6 | 6
Completed | 6 | 6 | 6
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated set [TS]: All subjects who received at least one dose of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | BI 1467335: Tablets, Fasted/Solution, Fasted/Tablets, Fed | BI 1467335: Solution, Fasted/Tablets, Fed/Tablets, Fasted | BI 1467335: Tablets, Fed/Tablets, Fasted/Solution, Fasted | Total
Number analyzed (Participants) | 6 | 6 | 6 | 18
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42.2 (12.2) | 45.7 (9.8) | 45.7 (6.3) | 44.5 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 6 | 6 | 6 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 6 | 5 | 6 | 17
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 6 | 6 | 6 | 18
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: AUC0-tz of BI 1467335
Description: This outcome measure presents AUC0-tz [area under the concentration-time curve of BI 1467335 in plasma over the time interval from 0 to the last quantifiable data point].
Time Frame: At -1:00h [hours (h): minutes (min)] before drug administration and at 0:15, 0:30, 0:45, 1:00, 1:15, 1:30, 1:45, 2:00, 2:30, 3:00, 4:00, 6:00, 8:00, 10:00, 12:00 and 24:00 h:min after drug administration.
Population: PharmacoKinetic Set [PKS]: This subject set included all subjects in the Treated Set [All subjects who received at least one dose of study medication] who provided at least one primary PK parameter that was not excluded due to a relevant protocol violation [PV] or non-evaluable plasma concentrations. One subject did not receive the dose in period 2 [Tablets, fed].
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomole*hour/Liter (nmol*h/L)
Groups:
- BI 1467335: Tablets, Fed: The subjects were administered BI 1467335 10 mg [2*5 mg] film-coated tablets orally in the fed state. The treatment duration was one day.
- BI 1467335: Tablets, Fasted: The subjects were administered BI 1467335 10 mg [2*5 mg] film-coated tablets in the fasted state orally with 240 mL of water after an overnight fast of at least 10h. The treatment duration was one day.
- BI 1467335: Solution, Fasted: The subjects were administered BI 1467335 10 mg oral solution in the fasted state orally with 240 mL of water after an overnight fast of at least 10h. The treatment duration was one day.
Arm/Group | BI 1467335: Tablets, Fed | BI 1467335: Tablets, Fasted | BI 1467335: Solution, Fasted
Number analyzed (Participants) | 17 | 18 | 18
nanomole*hour/Liter (nmol*h/L) | 3.90 (90.5) | 2.24 (101) | 2.49 (121)
Statistical Analysis 1: Comparison: BI 1467335: Tablets, Fasted vs BI 1467335: Solution, Fasted; The statistical model used for the analysis of the endpoint was an ANOVA [Analysis of Variance] model on the logarithmic scale. This model included effects accounting for the following sources of variation: 'sequence', 'subjects nested within sequences', 'period' and 'treatment'. The effect 'subjects within sequences' was considered as random, whereas the other effects were considered as fixed; Test type: Other; ANOVA; Ratio = 89.90, 90% CI 2-sided [73.304 to 110.25], Standard Deviation 36.0 — The estimated parameter was the adjusted geometric mean ratios [%] of BI 1467335: Tablets, fasted (numerator) and Solution, fasted (denominator). The Standard Deviation [SD] is the intra-individual geometric coefficient of variation [%]
Statistical Analysis 2: Comparison: BI 1467335: Tablets, Fed vs BI 1467335: Tablets, Fasted; [analysis description as in outcome 1, analysis 1]; Test type: Other; ANOVA; Ratio = 170.78, 90% CI 2-sided [139.85 to 208.54], Standard Deviation 33.9 — The estimated parameter was the adjusted geometric mean ratios [%] of BI 1467335: Tablets, fed (numerator) and Tablets, fasted (denominator). The parameter dispersion type [SD] is the intra-individual geometric coefficient of variation [%]

2. Primary Outcome: Cmax of BI 1467335
Description: This outcome measure presents the maximum measured concentration of BI 1467335 in plasma (Cmax of BI 1467335).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomole/Liter (nmol/L)
Arm/Group | BI 1467335: Tablets, Fed | BI 1467335: Tablets, Fasted | BI 1467335: Solution, Fasted
Number analyzed (Participants) | 17 | 18 | 18
nanomole/Liter (nmol/L) | 2.55 (120) | 1.85 (107) | 2.20 (126)
Statistical Analysis 1: Comparison: BI 1467335: Tablets, Fasted vs BI 1467335: Solution, Fasted; [analysis description as in outcome 1, analysis 1]; Test type: Other; ANOVA; Ratio = 84.17, 90% CI 2-sided [64.260 to 110.24], Standard Deviation 48.8 — The estimated parameter was the adjusted geometric mean ratios [%] of BI 1467335: Tablets, fasted (numerator) and Solution, fasted (denominator). The parameter dispersion type [SD] is the intra-individual geometric coefficient of variation [%]
Statistical Analysis 2: Comparison: BI 1467335: Tablets, Fed vs BI 1467335: Tablets, Fasted; [analysis description as in outcome 1, analysis 1]; Test type: Other; ANOVA; Ratio = 136.16, 90% CI 2-sided [99.885 to 185.61], Standard Deviation 54.8 — [estimate comment as in outcome 1, analysis 2]

ADVERSE EVENTS:
Time Frame: From the first day of study drug administration until 21 days after the first drug administration, up to 22 days.
Description: Treated set [TS]: All subjects who received at least one dose of study medication.
Arm/Group | BI 1467335: Tablets, Fasted | BI 1467335: Solution, Fasted | BI 1467335: Tablets, Fed
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/18 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18 | 0/17
Other Adverse Events (participants affected / at risk) | 2/18 | 5/18 | 4/17
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BI 1467335: Tablets, Fasted (N=18) | BI 1467335: Solution, Fasted (N=18) | BI 1467335: Tablets, Fed (N=17)
Bronchitis (Infections and infestations) | 0 | 0 | 1
Epididymitis (Infections and infestations) | 0 | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 1 | 1
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2016-10-12): https://cdn.clinicaltrials.gov/large-docs/91/NCT02999191/Prot_000.pdf
  • Statistical Analysis Plan (2017-05-15): https://cdn.clinicaltrials.gov/large-docs/91/NCT02999191/SAP_001.pdf